CLINICAL TRIAL: NCT03198208
Title: Effects of Intraoperative Fentanyl Dose on Postoperative Respiratory Complications
Brief Title: Intraoperative Fentanyl Dose on Respiratory Complications
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Matthias Eikermann, Associate Professor of Anaesthesia, Harvard Medical School; Clinical Director, Critical Care Division, Massachusetts General Hospital
Other Study IDs: 2017P000825
Record Dates: First submitted 2017-06-21; First posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Fentanyl; Opioid Use; Surgery; Respiratory Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reference group: No fentanyl dose administered during surgery
  Interventions: Drug: Fentanyl dose administration
- Comparative group: Fentanyl dose administered during surgery
  Interventions: Drug: Fentanyl dose administration

INTERVENTIONS:
Drug: Fentanyl dose administration

SUMMARY:
Fentanyl is the most commonly used opioid during anesthesia at Massachusetts General Hospital. Compared to other opioids, e.g. sulfentanil and remifentanil, fentanyl's pharmacokinetic properties are more problematic as the context sensitive half-time increases with duration of fentanyl infusion. This may lead to respiratory complications particularly in patients who receive fentanyl for surgical procedures of long duration. Considering the common use of fentanyl during surgery and its duration of action that is hard to predict during long surgical procedures, we will evaluate the association between intraoperative fentanyl dose and postoperative respiratory complications within 3 days of surgery.

DETAILED DESCRIPTION:
Our team has conducted a series of studies to define the optimal anesthesia plan that minimizes the risk of postoperative respiratory complications. Opioids are almost always used in the perioperative management of patients undergoing surgery during anesthesia. Intraoperatively they are administered to achieve adequate surgical conditions. Opioids are respiratory depressants. They decrease dose-dependently the drive to the respiratory pump muscles and upper airway dilator muscles, which leads to respiratory acidemia and hypercapnia. Fentanyl is the most commonly used opioid during anesthesia at MGH. Compared to other opioids, e.g. sulfentanil and remifentanil, fentanyls pharmacokinetic is more problematic as the context sensitive half-life increases with duration of fentanyl administration. This may lead to respiratory complications. Considering the common use of fentanyl during surgery and its duration of action that is hard to predict during long surgical procedures, we will evaluate the association between intraoperative fentanyl dose and postoperative respiratory complications within 3 days of surgery.

To account for other factors that may affect the incidence of postoperative respiratory complications, we included the following confounder model in all of our analyses:

* Gender
* Age
* BMI (body mass index)
* ASA status classification
* CCI (Charlson Comorbidity Index)
* Inhalational anesthetics as MAC
* Long lasting opioids as IV-morphine milligram equivalent including morphine, hydromorphone, methadone and sufentanil.
* Use of neuraxial anesthesia
* Intraoperative vasopressor dose
* Intraoperative NMBA (neuromuscular blocking agent) dose
* Intraoperative hypotension as number of minutes of an MAP (mean arterial pressure) <55 mmHG
* Duration of surgery
* Emergency status
* Intraoperative fluids
* PRBC (packed red blood cells) units
* Work RVU [relative value unit]
* Surgical service
* Admission type (ambulatory vs inpatient)
* SPORC (Score for Prediction of Postoperative Respiratory Complications)
* SPOSA (Score for Prediction of Obstructive Sleep Apnea)
* Inspiratory O2 - Fraction
* Protective ventilation (defined as PEEP=5 and plateau pressure between 0 and 16)
* Perioperative naloxone use
* Prescription of any of the following opioids within 90 days prior to surgery: oxycodone, codeine, hydrocodone, buprenorphine, butorphanol, opium, hydromorphone, fentanyl, meperidine, morphine, levorphanol, methadone, nalbuphine, tapentadol, oxymorphone, roxicodone, tramadol
* Code status (DNR)

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients at Massachusetts General Hospital and two affiliated community hospitals
* 18 years of age and older
* Only patients who required general anesthesia with an endotracheal tube for the surgical procedure and were extubated in the operating room at the end of the procedure.

Exclusion Criteria:

* Brain dead patients (ASA greater than 5)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with surgeries performed between 01/2007 and 12/2015 at Massachusetts General Hospital and two affiliated community hospitals.
Sampling Method: Probability Sample
Enrollment: 183396 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative respiratory complications | Between the day of surgery and the third day after surgery
  New postoperative respiratory complications occuring within 3 days after surgery

OTHER OUTCOMES:
Post-extubation desaturation | Immediately after endotracheal extubation at the end of surgery
  Oxygen saturation below 80% and 90% measured immediately after endotracheal extubation
Non-invasive ventilation | Between the day of surgery and the third day after surgery
  Incidence of non-invasive ventilation after surgery
ICU admission rate | Between day of surgery and hospital discharge, may be up to one year
  Admission to the ICU after surgery
Hospital length of stay | Number of days between day of hospital admission and hospital discharge, may be up to one year
  Total duration of hospitalized days
Total hospital costs | Between day of hospital admission and hospital discharge, may be up to one year
  Total costs for hospital stay
Wound infection | Between the day of surgery and 30 days after surgery
  Incidence of wound infection after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruscic KJ, Grabitz SD, Rudolph MI, Eikermann M. Prevention of respiratory complications of the surgical patient: actionable plan for continued process improvement. Curr Opin Anaesthesiol. 2017 Jun;30(3):399-408. doi: 10.1097/ACO.0000000000000465. PMID 28323670
- [Background] Thevathasan T, Shih SL, Safavi KC, Berger DL, Burns SM, Grabitz SD, Glidden RS, Zafonte RD, Eikermann M, Schneider JC. Association between intraoperative non-depolarising neuromuscular blocking agent dose and 30-day readmission after abdominal surgery. Br J Anaesth. 2017 Oct 1;119(4):595-605. doi: 10.1093/bja/aex240. PMID 29121289
- [Background] de Jong MAC, Ladha KS, Vidal Melo MF, Staehr-Rye AK, Bittner EA, Kurth T, Eikermann M. Differential Effects of Intraoperative Positive End-expiratory Pressure (PEEP) on Respiratory Outcome in Major Abdominal Surgery Versus Craniotomy. Ann Surg. 2016 Aug;264(2):362-369. doi: 10.1097/SLA.0000000000001499. PMID 26496082
- [Background] Ladha K, Vidal Melo MF, McLean DJ, Wanderer JP, Grabitz SD, Kurth T, Eikermann M. Intraoperative protective mechanical ventilation and risk of postoperative respiratory complications: hospital based registry study. BMJ. 2015 Jul 14;351:h3646. doi: 10.1136/bmj.h3646. PMID 26174419
- [Background] Shin CH, Grabitz SD, Timm FP, Mueller N, Chhangani K, Ladha K, Devine S, Kurth T, Eikermann M. Development and validation of a Score for Preoperative Prediction of Obstructive Sleep Apnea (SPOSA) and its perioperative outcomes. BMC Anesthesiol. 2017 May 30;17(1):71. doi: 10.1186/s12871-017-0361-z. PMID 28558716
- [Background] Brueckmann B, Villa-Uribe JL, Bateman BT, Grosse-Sundrup M, Hess DR, Schlett CL, Eikermann M. Development and validation of a score for prediction of postoperative respiratory complications. Anesthesiology. 2013 Jun;118(6):1276-85. doi: 10.1097/ALN.0b013e318293065c. PMID 23571640
- [Derived] Friedrich S, Raub D, Teja BJ, Neves SE, Thevathasan T, Houle TT, Eikermann M. Effects of low-dose intraoperative fentanyl on postoperative respiratory complication rate: a pre-specified, retrospective analysis. Br J Anaesth. 2019 Jun;122(6):e180-e188. doi: 10.1016/j.bja.2019.03.017. Epub 2019 Apr 11. PMID 30982564